CLINICAL TRIAL: NCT00180180
Title: Tumor Hypoxia of Head-and-neck Cancer Underwent Radiation Therapy Measured With F-18-FMISO
Status: Completed | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Principal Investigator, Jörg Kotzerke, Prof. Dr., Technische Universität Dresden
Other Study IDs: HNO-FMISO-FU
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Head and Neck Neoplasms
Keywords: head-and-neck cancer; radiation therapy; F-18-FMISO
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to describe the regional and global tumor hypoxia in head-and-neck cancer during percutaneous radiation therapy

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed head-and-neck cancer not curable by surgery
* Karnofsky > 70%
* tumor volume and localisation allow curative radiotherapy
* written consent

Exclusion Criteria:

* metastases
* earlier radiation therapy of head and neck
* pregnancy
* secondary malignancy excluding dermal carcinoma and Tis-carcinoma of cervix uteri
* psychiatric impairment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study includes consecutive patients from the Department of Radiooncology with head and neck cancer (HNC) intended for a curative chemoradiotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2006-07; Primary Completion 2017-03 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joerg Kotzerke, MD, Principal Investigator — Department of Nuclear Medicine
Locations (1):
- Department of Nuclear Medicine, Dresden, Germany